CLINICAL TRIAL: NCT06693817
Title: Advanced Wireless Sensors for Neonatal Care in the Delivery Room: the AWARD Prospective Multicenter International Study
Brief Title: Advanced Wireless Sensors for Neonatal Care in the Delivery Room
Acronym: AWARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guilherme Sant'Anna, MD (Other)
Collaborators: Federal University of Uberlandia (Other); University of Campinas, Brazil (Other); Sanatorio de la Trinidad Palermo (Unknown); Mbuya Nehanda Hospital Harare Zimbabwe (Unknown); Hopsital Central de Maputo, Mozambique (Unknown)
Responsible Party: Sponsor-Investigator, Guilherme Sant'Anna, MD, Senior Clinician Scientist, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AWARD Study
Record Dates: First submitted 2024-10-30; First posted 2024-11-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sudden Unexplained Infant Death; Apnea of Newborn; Newborn Morbidity; Newborn Asphyxia; Birth Outcome, Adverse; Birth Asphyxia; Pregnancy Related; Newborn; Vitality; ECG Electrode Site Reaction; Infant ALL; Infant Death; Infant, Newborn, Diseases; Infant Apnea; Infant Conditions; Parents; Delivery Problem for Fetus; Delivery Complication
Keywords: Delivery Room; Newborn; Neonatal Resuscitation; Wireless Technology; Vital Sign Monitoring; Sudden Unexplained Post-Natal Collapse; SUPC; Obstetrical Center; Obstetrics; Neonate; Birth; Birthing Center; C-Section; Vaginal Delivery; Sensors; Heart Rate (HR); Respiratory Rate (RR); Blood Oxygen Saturation (SpO2); Skin Temperature (Tskin); Pulse Rate (PR); International; Low-Income; Middle-Income; High-Income; Golden Hour; Post-Birth
MeSH Terms: conditions — Asphyxia Neonatorum; Pregnancy Complications; Infant Death; Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaginal Birth (Other): Wireless monitoring system placed first for vaginal birth. 15-20 minutes later, the wired monitoring system is placed. Both systems stay in place for 2 hours.
  Interventions: Device: Wireless skin sensors vital sign monitoring system; Device: Wired vital sign monitoring system
- C-Section Birth (Other): System placement randomized for C-section. One system placed first and the alternate placed immediately after. Both systems stay in place for 2 hours.
  Interventions: Device: Wireless skin sensors vital sign monitoring system; Device: Wired vital sign monitoring system

INTERVENTIONS:
Device: Wireless skin sensors vital sign monitoring system — The wireless monitoring system will be applied to the newborn and consist of a chest sensor (Anne Arc by Sibel Inc.) and a RAD-7 (Masimo)pulse oximeter limb sensor.
  Other Names: Anne Arc (Sibel Health Inc); Radical-7 (Masimo)
Device: Wired vital sign monitoring system — A standard ECG and SpO2 monitoring device will be applied suing the Infinity M540 monitor (Draeger, Germany). The chest sensor will be placed as per standard of care on the newborn's chest and abdomen, and the SpO2 sensor on their hands or feet.
  Other Names: Infinity M540 (Draeger)

SUMMARY:
The goals of this observational study is to assess whether a new advanced wireless skin sensor vital sign monitoring system can effectively monitor the vital signs of healthy newborn infants (≥ 35 weeks gestational age). The main aims of this Study are to:

1. Assess feasibility
2. Evaluate safety
3. Determine accuracy of the wireless monitoring system, compared to the standard of care wired vital sign monitoring system, immediately after delivery and for the first 2h of age in the obstetrical center under unsupervised parents' care. The newborn infants participating in the Study will have both vital sign monitoring systems placed on their chest and limb. Their vital signs will be monitored for 2h consecutively.

DETAILED DESCRIPTION:
When the transition from intrauterine to extrauterine life necessitates Neonatal Resuscitation, specialized monitoring of vital signs is required. Sudden Unexpected Postnatal Collapse (SUPC) is an apnea or cardiorespiratory failure occurring in otherwise healthy near-term or term neonates, usually in the first 48 hours of age, during the initial Kangaroo Mother Care (KMC) in the obstetrical center. SUPC carries a high morbidity and mortality rate. Approximately 10 million babies do not breathe immediately after birth, and 60% require basic resuscitation interventions. Sudden Unexpected Postnatal Collapse has been estimated to occur in 2.6-133 cases per 100.000 newborns and over 50% of the cases occur following accidental suffocation, which frequently goes unrecognised by parents in the obstetrical center during unsupervised KMC.

Current guidelines recommend monitoring of heart rate (HR), oxygen saturation (SpO2), and skin temperature (Tskin) during neonatal resuscitation. This is usually achieved by using wired electrodes and sensors that require expensive and large base units attached to a power supply. SUPC is a rare but largely preventable cause of neonatal mortality that deserves particular attention. Better resuscitation and prevention of SUPC might be achieved by continuous non-intrusive monitoring of vital signs immediately after delivery and while in the obstetrical center.

This research will address a very important gap in care; the need for safe and accurate advanced, non-invasive, and non-intrusive wireless technologies for monitoring of vital signs immediately after birth and during the immediate postnatal care, potentially preventing cases of SUPC while in the obstetrical center.

Reliable and low-cost wireless monitoring that could be used immediately after delivery would promote widespread adoption of neonatal resuscitation recommendations in low and middle income countries, improve detection of vital signs quickly after delivery and during early unsupervised KMC, and optimize neonatal care in the obstetrical centers or during hospital stay, to prevent cases of SUPC and its associated high mortality.

ELIGIBILITY:
Inclusion criteria:

1. Newborns ≥35 weeks (gestational age)
2. Newborns determined to be clinically stable at delivery
3. Newborns with no skin abnormalities

Exclusion criteria:

1. Newborns ≤ 35 weeks (gestational age)
2. Newborns determined to not be clinically stable at delivery
3. Newborns with Skin abnormalities

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using a wireless monitoring system immediately after delivery for HR. | 6 months
  Percentage of time for which heart rate (HR) is displayed.
Feasibility of using a wireless monitoring system immediately after delivery for RR. | 6 months
  Percentage of time for which respiratory rate (RR) is displayed.
Feasibility of using a wireless monitoring system immediately after delivery for SpO2. | 6 months
  Percentage of time for which blood oxygen saturation (SpO2) is displayed.
Feasibility of using a wireless monitoring system immediately after delivery for Tskin | 6 months
  Percentage of time for which skin temperature (Tskin) is displayed.
Feasibility of using a wireless monitoring system immediately after delivery - Gap occurence | 6 months
  Occurrence of gaps in signal detection/recordings (% and length in seconds).
Feasibility of using a wireless monitoring system immediately after delivery - Gap causes | 6 months
  Causes of the gaps in signal detection/recordings.
Feasibility of using a wireless monitoring system immediately after delivery - User satisfaction | 6 months
  Descriptive analysis of user surveys and their satisfaction with the wireless system.
Safety of using a wireless system immediately after delivery - skin score | 6 months
  Skin score (Neonatal Skin Condition Score) to be determined by a blinded dermatologist using de-identified pictures of the skin after removal of the sensors of each system. A "perfect" score using the NSCS is 3; the worst score is 9.
Safety of using a wireless system immediately after delivery - pain scale | 6 months
  Pain scale (Neonatal Infant Pain Scale) to assess any discomfort or pain during the removal of the sensors, with higher scores indicating greater pain.
Safety of using a wireless system immediately after delivery - clinical event discrepancies | 6 months
  Clinically significant events detected by the wired system (HR < 100 bpm or SpO2 < 80%) but missed by the wireless system.
Assess the accuracy of this wireless system - correlation coefficient. | 6 months
  Measuring HR, RR, SpO2 and Tskin signals compared with the "standard of care" wired system - Correlation coefficient
Assess the accuracy of this wireless system - slope | 6 months
  Measuring HR, RR, SpO2 and Tskin signals compared with the "standard of care" wired system - Slop
Assess the accuracy of this wireless system - variance accounted for | 6 months
  Measuring HR, RR, SpO2 and Tskin signals compared with the "standard of care" wired system - Variance accounted for
Assess the accuracy of this wireless system - bias. | 6 months
  Measuring HR, RR, SpO2 and Tskin signals compared with the "standard of care" wired system - Bias

SECONDARY OUTCOMES:
Time between sensors placement and data display (seconds) | 6 months
  To determine the time (seconds)between sensors placement and data display for each system (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Sant'Anna, MD, PhD, Principal Investigator — The Research institute of the McGill University Health Centre
Locations (7):
- Hospitals Sanatorio Trinidad Palermo, Buenos Aires, Argentina
- Brazil (2):
  - Hospital de Clínicas de Uberlândia, Umuarama, Minas Gerais
  - ii. Hospital da Mulher Jose Aristodemo Pinotti State University of Campinas -CAISM, São Paulo
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- Maputo Central Hospital, Maputo, Mozambique
- Mbuya Nehanda Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No